CLINICAL TRIAL: NCT01568151
Title: Testing Interventions to Motivate and Educate
Acronym: TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Electra Paskett, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: TIME; 1R01CA116487 (NIH); OSU 08073 (Other: Ohio State University)
Record Dates: First submitted 2012-03-19; First posted 2012-04-02 (Estimated); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Screening; Education; Testing
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Clinics (Active Comparator): Subjects recruited at the Intervention Clinics will first be provided with Clinic-directed interventions(Clinic-directed intervention program)including: 1)provider-directed interventions; 2)office-based systems; and 3) waiting room materials. If the subjects have not undergone colorectal cancer screening after 12 months, they will be provided with an individual patient-directed program consisting of the following stepped interventions: 1) tailored physician letter, easy-to-read educational materials, and an fecal occult blood test (FOBT)information sheet and card; 2) telephone counseling for those who do not respond to the letter; and 3) home visits by lay health advisors for those who do not respond to the letter or phone counseling.
  Interventions: Behavioral: Clinic-directed intervention program; Behavioral: Individual Patient-Directed Program
- Usual Care Clinics (No Intervention): Subjects recruited at the Usual Care Clinics (Control Clinics) will not receive any study intervention. The results of how many subjects undergo colorectal cancer screening at the Usual Care Clinics will be compared to the number that undergo colorectal cancer screening at the Intervention Clinics.

INTERVENTIONS:
Behavioral: Clinic-directed intervention program — Clinic-directed intervention program: Subjects recruited at the Intervention Clinics will first be provided with Clinic-directed interventions including: 1)provider-directed interventions (computerized case-based education, evidence-based guidelines, ask the expert; 2)office-based systems (risk assessment forms, procedure monitoring, follow-up protocol, audit with feedback, chart reminders); and 3) waiting room materials.
  Arms: Intervention Clinics
Behavioral: Individual Patient-Directed Program — If the subjects have not undergone colorectal cancer screening within 12 months of receiving the clinic-directed program, they will be provided with an individual patient-directed program consisting of the following stepped interventions: 1) tailored physician letter, easy-to-read educational materials, and an fecal occult blood test (FOBT)information sheet and card; 2) telephone counseling for those who do not respond to the letter; and 3) home visits by lay health advisors for those who do not respond to the letter or phone counseling.
  Arms: Intervention Clinics

SUMMARY:
This study is being done to see if teaching physicians and people who are at least 50 years old and have not been screened within guidelines for colorectal cancer about the importance of colorectal cancer screening will increase screenings for colorectal cancer. The researchers want to understand what ways will work best to motivate and educate both patients and the doctors and nurses who care for them.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third leading type of cancer and the third leading cause of cancer death in the United States. This study focuses on improving CRC screening in The Ohio State University Primary Care Network (OSUPCN). Ohio has higher than average rates of CRC mortality compared to the rest of the US. The study population for this study will also include minority and older individuals as these groups have higher CRC incidence and mortality rates.

The goal of this study is to test a program to improve CRC screening among male and female patients over the age of 50 in 10 primary care clinics. This study will use physician surveys, focus groups and a community advisory board to finalize the content of the interventions. Five theoretical models form the theoretical framework of the study - the health belief model, social networking, minority health communications model, PEN III, and the transtheoretical model. The interventions will be directed at the clinic and patient levels, and will be tested in a randomized design. Five clinics will receive the clinic plus patient-directed interventions and 5 clinics will be randomized to usual care. The clinic intervention will consist of provider, system and waiting room activities. The individual-directed intervention will include three stepped stages for patients who have not yet been screened: (1) a tailored physician letter, easy-to-read educational materials about CRC and an FOBT information sheet and card; (2) follow-up telephone barriers counseling for patients who do not complete CRC screening after receiving the letter; and (3) in person home visits by lay health advisors (LHA) for those who do not complete CRC screening after receiving the first two interventions. Research staff will conduct a process evaluation of the interventions to identify problems in implementing them and determine the extent to which each of the components is successfully carried out. They will also examine how components of the intervention relate to the theoretical frameworks used to motivate CRC screening completion. If successful, this program can easily be adapted for use by primary care practices and clinics to improve CRC screening.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* No prior history of familial/hereditary cancer syndrome (e.g. hereditary non-polyposis colon cancer), polyps, or inflammatory bowel disease (e.g. Crohn's disease)
* Have a current phone number
* Have had 2 or more visits to the Family Practice or General Internal Medicine Clinics in the past 2 years
* Have a current address in records and no definite plans to move within the next year
* Be at average risk for colorectal cancer
* Be in good health as judged by their primary care doctor
* Not be over the age of 85

Exclusion Criteria:

* Less than 50 years old
* Greater than 85 years old
* History of familial/hereditary cancer syndrome, polyps, or Crohn's disease
* History of contraindications to colorectal cancer screening, such as congenital heart failure, renal failure, dementia

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2009-04; Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who undergo colorectal screening because of interventions | Up to 3 and a half years
  The effectiveness of clinic-directed interventions in encouraging subjects to undergo colorectal cancer screening in the 5 intervention clinics in the first 12 months will be assessed. The subjects who did not undergo colorectal cancer screening during that year will then undergo patient-directed intervention for up to a year. The effectiveness of both of these types of intervention will be compared to the control clinics where there is no intervention.

SECONDARY OUTCOMES:
Number of problems associated with intervention program | Up to 3 and half years
  Conduct a process evaluation of the intervention program to identify problems experienced in implementing it. Process evaluation questions will be part of follow-up surveys that the participants complete. Responses will be analyzed by staff to determine intervention program concerns.

CONTACTS AND LOCATIONS:
Overall Officials: Electra D. Paskett, PhD, Principal Investigator — The Ohio State University Comprehensive Cancer Center
Locations (1):
- The Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murray DM, Katz ML, Post DM, Pennell ML, Young GS, Tatum CM, Paskett ED. Enhancing cancer screening in primary care: rationale, design, analysis plan, and recruitment results. Contemp Clin Trials. 2013 Mar;34(2):356-63. doi: 10.1016/j.cct.2013.01.003. Epub 2013 Jan 26. PMID 23357561
- See also: Jamesline — http://cancer.osu.edu